CLINICAL TRIAL: NCT02468232
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of LCZ696 Compared to Enalapril on Morbidity and Mortality in Japanese Patients With Chronic Heart Failure and Reduced Ejection Fraction.
Brief Title: Study of Efficacy and Safety of LCZ696 in Japanese Patients With Chronic Heart Failure and Reduced Ejection Fraction
Acronym: PARALLEL-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696B1301
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HF-rEF)
Keywords: chronic heart failure; cardiovascular death; hospitalization; outcome study; worsening heart failure; NT-proBNP; NYHA; KCCQ; HF-rEF
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCZ696 (Experimental): Before randomization, all patients received 2 week LCZ696 50 mg twice daily (b.i.d) as single blind run-in active treatment epoch. In double blind epoch, randomized patients in this arm started with 100 mg twice daily (b.i.d.) for 4 weeks. Patients were then up-titrated to 200 mg b.i.d. at week 4 if they were tolerant to 100 mg b.i.d. Total duration of treatment was up to approximately 40 months.
  Interventions: Drug: LCZ696; Drug: Placebo to Enalapril
- Enalapril (Active Comparator): Before randomization, all patients received 2 week LCZ696 50 mg twice daily (b.i.d) as single blind run-in active treatment epoch. In double blind period, all randomized patients in this arm received enalapril 5mg twice daily (b.i.d.) for 4 weeks. Patients were then up-titrated to 10 mg b.i.d. at week 4 if they were tolerant to 5 mg b.i.d. Total duration of treatment was up to approximately 40 months.
  Interventions: Drug: Enalapril; Drug: Placebo to LCZ696

INTERVENTIONS:
Drug: LCZ696 — The target dose during the study was LCZ696 200 mg bid given orally. LCZ696 was supplied as 50 mg, 100 mg and 200 mg film-coated tablets.
  Arms: LCZ696
Drug: Enalapril — The target dose during the study was enalapril 10 mg bid given orally. Enalapril was provided as 2.5 mg, 5 mg, and 10 mg tablets.
  Arms: Enalapril
Drug: Placebo to LCZ696 — LCZ696 Placebo 50 mg, 100 mg and 200 mg film-coated tablets
  Arms: Enalapril
Drug: Placebo to Enalapril — Enalapril Placebo 2.5 mg, 5 mg and 10 mg tablets
  Arms: LCZ696

SUMMARY:
The purpose of this study was to assess the effect of LCZ696 at a target dose of 200 mg b.i.d. compared to enalapril 10 mg b.i.d., in addition to the background heart failure (HF) treatment, on delaying time to first occurrence of either cardiovascular (CV) death or HF hospitalization events in Japanese patients with stable chronic heart failure (CHF), New York Heart Association (NYHA) classes II-IV and reduced ejection fraction (left ventricular ejection fraction (LVEF) ≤ 35%).

DETAILED DESCRIPTION:
The study consisted of two parts: the core part and the Open label extension (OLE) epoch.

The core part of this study was a multicenter, randomized, double-blind, double-dummy, parallel-group, active-controlled study to assess the effect of LCZ696 at a target dose of 200 mg b.i.d. and enalapril 10 mg b.i.d. on CV mortality and morbidity reduction in Japanese HF patients with reduced ejection fraction. Patients who met the eligibility criteria at screening entered a 2 week, single-blind, active treatment run-in epoch in which they received LCZ696 50 mg b.i.d. Patients who tolerated LCZ696 50 mg b.i.d. for 2 weeks were randomized in a 1:1 ratio to receive LCZ696 100 mg b.i.d. or enalapril 5 mg b.i.d. for 4 weeks during the double-blind treatment epoch. The patient randomization was stratified by using NT-proBNP measured at the screening visit as a stratification factor. The patients were then titrated up to the target dose of LCZ696 200 mg b.i.d. or enalapril 10 mg b.i.d. if they tolerated 4 weeks treatment of LCZ696 100 mg b.i.d. or enalapril 5 mg b.i.d. Dose adjustment (LCZ696 50-100 mg b.i.d. & enalapril 2.5-5 mg b.i.d.) was permitted if not tolerated at the target dose of study drugs during the double-blind treatment epoch.

This was an event-driven study in which subjects remained on the study (regardless of whether receiving investigational medications) until the projected number of patients with primary events (approximately 57 events) had been reached.

The Open label extension (OLE) epoch was conducted following the completion of the core part, with the aim to provide access to LCZ696 for eligible subjects until the marketed product was available in Japan or 2 years from the date of the first subject enrolled in the OLE epoch, whichever occurred first, and also to obtain the safety and tolerability data of long-term treatment with LCZ696.

Upon completion of the core part, the eligibility of the subjects to enter the OLE epoch was assessed by the investigator at OLE baseline (Visit 301), which occurred on the same day as the end of study (EOS) visit of the core part (Visit 299). At this visit, subjects were switched to open-label LCZ696.

At Visit 302 (2 to 4 weeks after Visit 301), subjects who tolerated the open-label LCZ696 and met the safety monitoring criteria were up-titrated to the next higher level of daily dose. Thereafter, subject visits occurred at 8 weeks, and then every 4 months until EOS visit for OLE epoch.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Outpatients with a diagnosis of CHF NYHA class II-IV and reduced ejection fraction:
* LVEF ≤ 35% at Visit 1 (any local measurement, made within the past 6 months using echocardiography, MUGA, CT scanning, MRI or ventricular angiography is also acceptable, provided no subsequent measurement above 35%)
* NT-proBNP ≥ 600 pg/ml at Visit 1 OR NT-proBNP ≥ 400 pg/ml at Visit 1 and a hospitalization for HF within the last 12 months (according to central laboratory measurements)
* Patients must be on an ACEI or an ARB at a stable dose for at least 4 weeks before Visit 1.
* Patients must be treated with a β-blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks prior to Visit 1 (reason should be documented if patients reported contraindications or intolerance).
* An aldosterone antagonist should also be considered in all patients, taking account of renal function, serum potassium and tolerability. If given, the dose of aldosterone antagonist should be optimized according to guideline recommendations and patient tolerability, and should be stable for at least 4 weeks prior to Visit 1. Other evidence-based therapy for HF should also be considered e.g. cardiac resynchronization therapy and an implantable cardioverter-defibrillator in selected patients, as recommended by guidelines.

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes, ACEIs, ARBs, NEP inhibitors as well as known or suspected contraindications to the study drugs.
* Previous documented history of intolerance to ACEIs or ARBs.
* Known history of angioedema.
* Requirement of treatment with both ACEIs and ARBs.
* Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy).
* Symptomatic hypotension and/or a SBP < 100 mmHg at screening or < 95 mmHg at the end of run-in.
* Estimated GFR < 30 mL/min/1.73 m2 as measured by the Japanese formula at screening, or the end of run-in or > 35% decline in eGFR between screening and end of run-in (according to local measurements).
* Serum potassium > 5.2 mmol/L (mEq/L) at screening or > 5.4 mmol/L (mEq/L) at the end of run-in (according to local measurements).
* Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major CV surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within the 3 months prior to Visit 1.
* Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months prior to Visit 1.
* Symptomatic bradycardia or second (except asymptomatic Wenckebach block) or third degree heart block without a pacemaker.
* Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
* Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
* Presence of bilateral renal artery stenosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2021-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Japan (46):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Hatsukaichi, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Otaru, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Uji, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Miyazaki, Miyazaki
  - Novartis Investigative Site, Saku, Nagano
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Yonago, Tottori
  - Novartis Investigative Site, Shūnan, Yamaguchi
  - Novartis Investigative Site, Kofu, Yamanashi
  - Novartis Investigative Site, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was estimated that approximately 370 patients would be screened in order to randomize 220 patients (110 patients in each arm), as the screen or run-in failure rate was anticipated to be approximately 40%. It was anticipated that approximately 180 subjects would complete the core part of the study & majority of them would be enrolled into the open-label extension (OLE).
Pre-assignment Details: Overall, 307 patients were screened, and 71 patients discontinued prior to the screening epoch completion. Thus, 236 patients entered the run-in epoch, with 11 patients being run-in failures.
Groups:
- LCZ696 (Core) OLE Epoch: The patients who received LCZ696 in the core part of the study and continued to receive LCZ696 in the open-label extension (OLE) are referred to as LCZ (core) group. These patients received open-label LCZ696 in the OLE phase.
- Enalapril (Core) OLE Epoch: The subjects who received enalapril in the core part and then switched to LCZ696 in the OLE are referred to as ENA (core) group. These patients switched from enalapril and received open-label LCZ696 in the OLE phase.
Period: Core Part of Study
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Started (Started = Enrolled in Core) | 112 | 113 | 0 | 0
Randomized Patients | 112 | 113 | 0 | 0
Mis-randomized Patients | 1 | 1 | 0 | 0
Discont. From Randomized Treatment (Rand. Set) | 21 | 19 | 0 | 0
Discont. From Rand. Treatment (Full Analysis Set) | 20 | 18 | 0 | 0
Completed (Completed = Completed Core) | 91 | 94 | 0 | 0
Not Completed | 21 | 19 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 20 | 17 | 0 | 0
Not completed — Technical Problems | 1 | 1 | 0 | 0
Period: OLE Part of Study
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Started | 0 | 0 | 79 | 71
Completed | 0 | 0 | 65 | 59
Not Completed | 0 | 0 | 14 | 12
Not completed — Adverse Event | 0 | 0 | 4 | 5
Not completed — Death | 0 | 0 | 4 | 2
Not completed — Physician Decision | 0 | 0 | 4 | 0
Not completed — Subject/Guardian decision | 0 | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consists of all randomized patients with the exception for those patients who have not been qualified for randomization (mis-randomized) and have not received investigational drug, but have been inadvertently randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch | Total
Number analyzed (Participants) | 111 | 112 | 0 | 0 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.97 (9.717) | 66.70 (10.938) |  |  | 67.83 (10.388)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 |  |  | 31
  Male | 96 | 96 |  |  | 192
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 111 | 112 |  |  | 223

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had CEC (Clinical Endpoint Committee) Confirmed Composite Endpoints
Description: Composite endpoint is defined as either cardiovascular (CV) death or heart failure (HF) hospitalization in Japanese patients with chronic heart failure (CHF) and reduced ejection fraction. The composite endpoint events occurred on and after End-of-study (EOS) declaration were reported by investigators but those events were not required to be adjudicated by Clinical Endpoint Committee (CEC) and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: FAS consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants
  Primary composite | 30 | 28 | 0 | 0
  Cardiovascular (CV) Death | 13 | 11 | 0 | 0
  1st heart failure (HF) Hospitalization | 25 | 20 | 0 | 0

2. Primary Outcome: Exposure-adjusted Incident Rate (EAIR) of CEC Confirmed Composite Endpoints
Description: Composite endpoint is defined as either cardiovascular (CV) death or heart failure (HF) hospitalization in Japanese patients with chronic heart failure (CHF) and reduced ejection fraction. EAIR = n/T where n = Total number of events included in the analysis. T (100 patient years) = total up-to-event/censoring duration-time summarized over participants in the respective treatment group. The composite endpoint events occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 patient-years
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Events per 100 patient-years
  Primary composite | 11.376 [7.676 to 16.240] | 10.497 [6.975 to 15.170] |  |
  Cardiovascular (CV) Death | 4.410 [2.348 to 7.542] | 3.734 [1.864 to 6.681] |  |
  1st heart failure (HF) Hospitalization | 9.480 [6.135 to 13.995] | 7.498 [4.580 to 11.579] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; For Primary Composite; Test type: Superiority; p = 0.6260, Regression, Cox; Hazard Ratio (HR) = 1.0881, 95% CI 2-sided [0.6501 to 1.8212]
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; For CV Death; Test type: Superiority; p = 0.6493, Regression, Cox; Hazard Ratio (HR) = 1.1701, 95% CI 2-sided [0.5242 to 2.6122]
Statistical Analysis 3: Comparison: LCZ696 vs Enalapril; For 1st HF Hospitalization; Test type: Superiority; p = 0.7851, Regression, Cox; Hazard Ratio (HR) = 1.2673, 95% CI 2-sided [0.7039 to 2.2818]

3. Secondary Outcome: Key Secondary: Change From Baseline to the Pre-defined Time-points in Log-transformed Concentration of N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP is small protein produced in large amounts when the heart senses it needs to work harder, such as in heart failure. Change from baseline to the pre-defined time-points in logarithmic scale were analyzed using a repeated measures ANCOVA model with treatment, the stratification factor screening NT-proBNP classification recorded in the Interactive Web Response System (IWRS), visit and treatment-by-visit interaction as fixed effect factors and the logarithmic baseline biomarker value as a covariate, with a common unstructured covariance matrix among visits for each treatment. The analysis is using all available data up to month 6 based on likelihood method with an assumption of missing at random (MAR) for missing data.
  This record summarizes the estimates of ratio Post-baseline /Baseline NT-proBNP.
Time Frame: Baseline, Weeks 4, 8 and Month 6
Population: FAS consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study.
  This analysis is a longitudinal data analysis and all available data up to month 6 for each patient was used. Number of participants at each post-time point indicates the number of patients who have both baseline and post-time point values.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
ratio
  Week 4 (n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Week 4 (n = 111, 110, 0, 0) | 0.7672 [0.6988 to 0.8423] | 0.8862 [0.8071 to 0.9731] |  |
  Week 8 (n = 111, 108, 0, 0): number analyzed (Participants) | 111 | 108 | 0 | 0
  Week 8 (n = 111, 108, 0, 0) | 0.7798 [0.7123 to 0.8537] | 0.9134 [0.8339 to 1.0004] |  |
  Month 6 (n= 110, 106, 0, 0): number analyzed (Participants) | 110 | 106 | 0 | 0
  Month 6 (n= 110, 106, 0, 0) | 0.6947 [0.6210 to 0.7771] | 0.8564 [0.7646 to 0.9592] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Week 4 analysis; Test type: Superiority; p = 0.0326, ANCOVA — Indicates statistical significance (2-sided) with an alpha level of 0.05; Repeated measure ANCOVA model; LSM of ratio = 0.8657, 95% CI 2-sided [0.7585 to 0.9880]
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; Week 8 analysis; Test type: Superiority; p = 0.0161, ANCOVA — Indicates statistical significance (2-sided) with an alpha level of 0.05; Repeated measure ANCOVA model; LSM of ratio = 0.8538, 95% CI 2-sided [0.7509 to 0.9708]
Statistical Analysis 3: Comparison: LCZ696 vs Enalapril; Month 6 analysis; Test type: Superiority; p = 0.0104, ANCOVA — Indicates statistical significance (2-sided) with an alpha level of 0.05; Repeated measure of ANCOVA model; LSM of ratio = 0.8112, 95% CI 2-sided [0.6916 to 0.9514]

4. Secondary Outcome: Key Secondary: Number of Participants With CEC-confirmed First Triple Composite Endpoint (Cardiovascular (CV) Death, Heart Failure (HF) Hospitalization, or Worsening of HF in Outpatients)
Description: Composite endpoint is defined as either cardiovascular (CV) death or heart failure (HF) hospitalization in Japanese patients with chronic heart failure (CHF) and reduced ejection fraction. Worsening HF defined as: worsening signs and symptoms of HF requiring addition of a new drug for HF treatment, initiation of IV treatment, increase of diuretic dose for persistent use for ≥4 consecutive weeks, or institution of mechanical or circulatory support such as mechanical ventilation, ultrafiltration, hemodialysis, intra-aortic balloon pump or ventricular assist device. The composite endpoint events occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants
  First triple composite endpoint | 37 | 37 |  |
  CV death | 13 | 11 |  |
  First HF Hospitalization | 25 | 20 |  |
  First worsening of HF in outpatient | 12 | 14 |  |

5. Secondary Outcome: Key Secondary: EAIR of CEC-confirmed First Triple Composite Endpoint (Cardiovascular (CV) Death, Heart Failure (HF) Hospitalization, or Worsening of HF in Outpatients)
Description: Worsening HF defined as: worsening signs and symptoms of HF requiring addition of a new drug for HF treatment, initiation of IV treatment, increase of diuretic dose for persistent use for ≥4 consecutive weeks, or institution of mechanical or circulatory support such as mechanical ventilation, ultrafiltration, hemodialysis, intra-aortic balloon pump or ventricular assist device.
  EAIR(Exposure-adjusted incidence rate per 100 patient years)= n/T:
  n: Total number of events included in the analysis. T(100 patient years): total up-to-event/censoring duration-time summarized over patients in the respective treatment group. The composite endpoint events occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 patient-years
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Events per 100 patient-years
  First triple composite endpoint | 14.725 [10.368 to 20.297] | 14.479 [10.194 to 19.957] |  |
  CV death | 4.410 [2.348 to 7.542] | 3.734 [1.864 to 6.681] |  |
  First HF Hospitalization | 9.480 [6.135 to 13.995] | 7.498 [4.580 to 11.579] |  |
  First worsening of HF in outpatient | 4.372 [2.259 to 7.638] | 5.095 [2.786 to 8.549] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; First triple composite endpoint; Test type: Superiority; p = 0.5406, Regression, Cox; Hazard Ratio (HR) = 1.0240, 95% CI 2-sided [0.6492 to 1.6152]
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; CV health; Test type: Superiority; p = 0.6493, Regression, Cox; Hazard Ratio (HR) = 1.1701, 95% CI 2-sided [0.5242 to 2.6122]
Statistical Analysis 3: Comparison: LCZ696 vs Enalapril; First worsening of HF in outpatient; Test type: Superiority; p = 0.3448, Regression, Cox; Hazard Ratio (HR) = 0.8546, 95% CI 2-sided [0.3952 to 1.8479]

6. Secondary Outcome: Key Secondary: Number of Participants by Changes in New York Heart Association (NYHA) Classification From Baseline at Predefined Timepoints
Description: NYHA classification is a subjective physician's assessment of heart failure patient's functional capacity and symptomatic status.
  Class I - No limitation of physical activity. Class II - Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). Class III - Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. Class IV - Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  The NYHA class change was analyzed as a three category ordinal variable with levels: "improved", "unchanged", and "worsened", defined by at least one class improvement, no change, at least one class worsening, in NYHA class, respectively. NYHA class after patients who died was categorized into "worsened".
Time Frame: Baseline, Weeks 4, 8 and Month 6
Population: FAS consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study. Number of participants at post-time point (i.e., n) indicates the number of patients who have post-time point values.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants
  Week 4 Improved (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 4 Improved (n = 111, 111, 0, 0) | 8 | 10 |  |
  Week 4 Unchanged (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 4 Unchanged (n = 111, 111, 0, 0) | 102 | 96 |  |
  Week 4 Worsened (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 4 Worsened (n = 111, 111, 0, 0) | 1 | 5 |  |
  Week 8 Improved (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 8 Improved (n = 111, 111, 0, 0) | 15 | 12 |  |
  Week 8 Unchanged (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 8 Unchanged (n = 111, 111, 0, 0) | 95 | 93 |  |
  Week 8 Worsened (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 8 Worsened (n = 111, 111, 0, 0) | 1 | 6 |  |
  Month 6 Improved (n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Month 6 Improved (n = 111, 110, 0, 0) | 19 | 18 |  |
  Month 6 Unchanged (n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Month 6 Unchanged (n = 111, 110, 0, 0) | 91 | 84 |  |
  Month 6 Worsened (n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Month 6 Worsened (n = 111, 110, 0, 0) | 1 | 8 |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Week 4 analysis; Test type: Superiority; p = 0.7115, Cochran-Mantel-Haenszel; based on modified ridit scores
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; Week 8 analysis; Test type: Superiority; p = 0.1752, Cochran-Mantel-Haenszel; based on modified ridit scores
Statistical Analysis 3: Comparison: LCZ696 vs Enalapril; Month 6 analysis; Test type: Superiority; p = 0.2688, Cochran-Mantel-Haenszel; based on modified ridit scores

7. Secondary Outcome: Key Secondary: Change From Baseline in Clinical Summary Score for Heart Failure Symptoms and Physical Limitations Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ).
Description: The KCCQ is a self-administered questionnaire and requires, on average, 4-6 minutes to complete. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and Quality of Life (QoL), each with different Likert scaling wording, including limitations, frequency, bother, change in condition, understanding, etc. The clinical summary score is a mean of the physical limitation and total symptom scores. The total symptom score is the mean of the symptom frequency and symptom burden scores. Each scale score (the physical limitation, symptom frequency or symptom burden) is calculated as the mean of its item scores and transformed to a 0-100 scale, with higher score indicating higher level of functioning. A score of 100 represents perfect health whereas a score of 0 represents dead. A change of 5 points on the scale scores, either as a group mean difference or an intra-individual change appears to be clinically significant.
Time Frame: Baseline, Week 8 and Month 6
Population: FAS consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study. FAS included all patients with at least one KCCQ data. This is a longitudinal data analysis and all available data for each patient was used. Number of patients at each post-time point (n) indicates the number of patients who have both baseline and post-time point values.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
scores on a scale
  Week 8 (n = 111, 111, 0, 0): number analyzed (Participants) | 111 | 111 | 0 | 0
  Week 8 (n = 111, 111, 0, 0) | -0.0491 (1.3522) | -2.5946 (1.3504) |  |
  Month 6 (n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Month 6 (n = 111, 110, 0, 0) | -2.2216 (1.5898) | -3.4910 (1.5911) |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Week 8 analysis; Test type: Superiority; p = 0.1854, ANCOVA; Repeated measure ANCOVA model; LSM of difference = 2.5455, 95% CI 2-sided [-1.2306 to 6.3216]
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; Month 6 analysis; Test type: Superiority; p = 0.5737, ANCOVA; Repeated measure ANCOVA model; LSM of difference = 1.2695, 95% CI 2-sided [-3.1715 to 5.7104]

8. Secondary Outcome: Total Number of CEC Confirmed Composite of CV Death and Total (First and Recurrent) HF Hospitalizations for Heart Failure
Description: Total number of CEC-confirmed CV death and total (first and recurrent) HF hospitalizations per patient was analyzed using the negative binomial regression model. CV deaths and HF hospitalizations occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up tp 40 months
Population: The Full Analysis Set (FAS) consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study.
Measure: Number (95% Confidence Interval); unit: Events per patient
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Events per patient | 0.1734 [0.1123 to 0.2680] | 0.1994 [0.1295 to 0.3070] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.6501, Negative binomial (NB) regression model; adjusted for treatment and stratification of screening NT-proBNP; rate ratio = 0.8699, 95% CI [0.4763 to 1.5887]

9. Secondary Outcome: Number of Participants by Changes in Clinical Composite Score (as Assessed by NYHA Classification and Patient Global Assessment) at Predefined Timepoints
Description: The global assessment was derived from the 7-category classification of the global assessment of disease activity to a three-category classification: Improved (Markedly improved; moderately improved), Unchanged (Slightly improved, unchanged, slightly worsened), and Worsened (Moderately worsened, markedly worsened).
  The clinical composite assessment was defined as follows:
  * Improved: 1) If NYHA class decreased at least one level and Global Assessment was not worse at the selected visit and there was no major AE up to the selected visit; or 2) Global assessment was improved and NYHA class did not increase at the selected visit, and there was no major AE up to the selected visit.
  * Worsened: 1) If NYHA class increased at the selected visit; or 2) Global Assessment was worse at the selected visit; or 3) experienced a major AE up to the selected visit.
  * Unchanged: If neither "Improved" nor "Worsened".
Time Frame: Baseline, Month 6
Population: The Full Analysis Set (FAS) consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study. Overall Number of Participants Analyzed' indicates the number of patients who have post-time point values.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 110 | 110 | 0 | 0
Participants
  Clinical composite assessment: Improved | 23 | 21 |  |
  Clinical composite assessment: Unchanged | 78 | 78 |  |
  Clinical composite assessment: Worsened | 9 | 11 |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.6211, Cochran-Mantel-Haenszel

10. Secondary Outcome: Number of Participants With All-cause Mortality
Description: The number of participants who died due to any cause. Deaths occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants | 19 | 16 |  |

11. Secondary Outcome: EAIR of All-cause Mortality
Description: EAIR (Exposure-adjusted incidence rate per 100 patient years)= n/T:
  n: Total number of events included in the analysis. T(100 patient years): total up-to-event/censoring duration-time summarized over patients in the respective treatment group. Deaths occurred on and after EOS declaration were reported by investigators but those events were not required to be adjudicated by CEC and not included in the efficacy analysis.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Events per 100 patient-years
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Events per 100 patient-years | 6.445 [3.881 to 10.065] | 5.431 [3.104 to 8.820] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.6955, Regression, Cox; Hazard Ratio (HR) = 1.1895, 95% CI 2-sided [0.6116 to 2.3134]

12. Secondary Outcome: Percentage of Participants Hospitalized
Description: Percentage of participants with hospitalized admissions
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants | 62 | 62 |  |

13. Secondary Outcome: Hospitalization Admissions Events Per-participant Per Year
Description: The number of hospital admission events per-participant per year was calculated as total number of hospital admission divided by total up-to-event/censoring duration-time summarized over patients.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Hospitalization admissions per year
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Hospitalization admissions per year | 0.5881 [0.4439 to 0.7792] | 0.5771 [0.4376 to 0.7610] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.9233, Negative binomial (NB) regression model; adjusted for treatment and stratification of screening NT-proBNP; Rate ratio = 1.0192, 95% CI 2-sided [0.6925 to 1.4999]

14. Secondary Outcome: Days in Intensive Care Unit (ICU) Per Participant Per Year
Description: The number of days in ICU per participant per year was calculated as total number of days in ICU divided by total up-to-event/censoring duration-time summarized over patients.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Days per year
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Days per year | 0.8542 [0.2662 to 2.7409] | 0.7943 [0.2929 to 2.1541] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.9272, Negative binomial (NB) regression model; adjusted for treatment and stratification of screening NT-proBNP; Rate ratio = 1.0754, 95% CI 2-sided [0.2264 to 5.1067]

15. Secondary Outcome: Percentage of Re-hospitalizations
Description: The percentage of participants who had re-hospitalizations.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Participants
  2 Events | 10 | 16 |  |
  3 Events | 12 | 4 |  |
  4 Events | 2 | 4 |  |
  >= 5 Events | 10 | 11 |  |

16. Secondary Outcome: Emergency Department/Urgent Care Facility Visits for HF Per Patient Per Year
Description: The number of emergency department/urgent care facility visits for HF per patient per year was calculated as total number of emergency department/urgent care facility visits for HF divided by total up-to-event/censoring duration-time summarized over patients.
Time Frame: up to 40 months
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Visits per year
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
Visits per year | 0.0533 [0.0277 to 0.1025] | 0.1183 [0.0667 to 0.2097] |  |
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.0697, Negative binomial (NB) regression model — Negative binomial (NB) regression model; adjusted for treatment and stratification of screening NT-proBNP; Rate ratio = 0.4504, 95% CI 2-sided [0.1902 to 1.0665]

17. Secondary Outcome: Change in Blood NT-proBNP From Baseline
Description: NT-proBNP is small protein produced in large amounts when the heart senses it needs to work harder, such as in heart failure. Mean change from baseline (post-baseline value - baseline value) in plasma NT-proBNP was caluculated.
Time Frame: Baseline, Weeks 2, 4, 8 and Month 6
Population: The Full Analysis Set (FAS) consists of all randomized patients with the exception for those patients who have not been qualified for randomization and have not received investigational drug, but have been inadvertently randomized into the study. Number of participants at each post-time point (i.e., n) indicates the number of patients who have both baseline and post-time point values.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
pg/mL
  Week 2 (n = 111, 108, 0, 0): number analyzed (Participants) | 111 | 108 | 0 | 0
  Week 2 (n = 111, 108, 0, 0) | -366.5766 (611.8846) | -86.2222 (1997.9885) |  |
  Week 4 ( n = 111, 110, 0, 0): number analyzed (Participants) | 111 | 110 | 0 | 0
  Week 4 ( n = 111, 110, 0, 0) | -233.9279 (725.9590) | -224.8545 (2023.1202) |  |
  Week 8 (n = 111, 108, 0, 0): number analyzed (Participants) | 111 | 108 | 0 | 0
  Week 8 (n = 111, 108, 0, 0) | -252.0090 (590.5862) | -234.2963 (1840.3993) |  |
  Month 6 (110, 106, 0, 0): number analyzed (Participants) | 110 | 106 | 0 | 0
  Month 6 (110, 106, 0, 0) | -327.5000 (731.9563) | -240.7264 (2041.3829) |  |

18. Secondary Outcome: Change in Procollagen Type III N-Terminal Propeptide From Baseline
Description: Procollagen Type III N-Terminal Propeptide (PIIINP) is a serum marker of collagen turnover, generated during the synthesis of type III collagen. Increased circulating PIIINP is a marker not only of muscle growth, but also of muscle repair and fibrosis. Mean change from baseline (post-baseline value - baseline value) in serum PIIINP was calculated.
Time Frame: Baseline and Month 18
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 103 | 100 | 0 | 0
ug/L | 0.2914 (1.9105) | -0.0583 (1.7774) |  |

19. Secondary Outcome: Changes in Urine Cyclic Guanosine 3',5'-Monophosphate (cGMP) From Baseline
Description: Urinary Cyclic GMP (cGMP) is a biomarker measured in the urine that reflects the activity of biomarkers such as BNP (Brain Natriuretic Peptide). First morning void (FMV) urine samples were collected. Mean change from baseline (post-baseline value - baseline value) in urine cGMP was calculated.
Time Frame: Baseline, Weeks 4, 8 and Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 111 | 112 | 0 | 0
nmol/L
  Week 4 (n = 110, 109, 0, 0): number analyzed (Participants) | 110 | 109 | 0 | 0
  Week 4 (n = 110, 109, 0, 0) | 556.3182 (663.8357) | -25.9725 (552.6414) |  |
  Week 8 (n = 111, 107, 0, 0): number analyzed (Participants) | 111 | 107 | 0 | 0
  Week 8 (n = 111, 107, 0, 0) | 587.4414 (886.4691) | -52.7944 (503.1090) |  |
  Month 6 (n = 110, 102, 0, 0): number analyzed (Participants) | 110 | 102 | 0 | 0
  Month 6 (n = 110, 102, 0, 0) | 507.9182 (1169.4057) | -41.9706 (512.6963) |  |

20. Secondary Outcome: Percentage of Participants Reaching Target Dose Level 3 at Week 8 and Maintained at Month 4 (Open Label Extension (OLE))
Description: The percentage of participants who reached target dose level (200 mg b.i.d.) at Week 8 and maintained at Month 4(OLE). This indicates how tolerabile to LCZ696 at target dose.
Time Frame: Month 4 of OLE
Population: FAS-Ext: The full analysis set for OLE epoch (FAS-Ext) included all subjects in the extension population who received at least one dose of the extension study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
Participants |  |  | 51 | 52

21. Secondary Outcome: Change in NYHA Classification From OLE Baseline (OLE)
Description: as for outcome 6
Time Frame: OLE Baseline, Month 12 (OLE)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 71 | 66
Participants
  Improved |  |  | 3 | 4
  Unchanged |  |  | 64 | 60
  Worsened |  |  | 4 | 2

22. Secondary Outcome: Change in Key Echocardiographic Parameters From OLE Baseline at Month 12 (OLE)
Description: Key echocardiographic parameters:
  LAVi- left atrial volume index, LVEDVi- left ventricular end diastolic volume index, LVESVi- left ventricular end systolic volume index.
  A two-dimensional and doppler echo examination was done to assess echo parameters. Mean changes from baseline (post-baseline value - baseline value) in each parameter were calculated. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 12 (OLE)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
mL/m^2
  LAVi (n = 0, 0, 67, 55): number analyzed (Participants) | 0 | 0 | 67 | 55
  LAVi (n = 0, 0, 67, 55) |  |  | -3.31 (11.679) | -1.47 (12.389)
  LVEDVi (n = 0, 0, 62, 53): number analyzed (Participants) | 0 | 0 | 62 | 53
  LVEDVi (n = 0, 0, 62, 53) |  |  | 2.54 (18.712) | 0.99 (25.919)
  LVESVi (n = 0, 0, 62, 53): number analyzed (Participants) | 0 | 0 | 62 | 53
  LVESVi (n = 0, 0, 62, 53) |  |  | -2.32 (14.801) | -2.65 (20.619)

23. Secondary Outcome: Change in Cardiac Measurements by Key Echocardiographic Parameter LVEF, From OLE Baseline at Month 12 (OLE)
Description: Key echocardiographic parameter:
  LVEF- left ventricular ejection fraction. LVEF is a measurement expressed as a percentage of how much blood the left ventricle pumps out with each contraction. Mean changes from baseline (post-baseline value - baseline value) in LVEF were calculated.
Time Frame: Baseline, Month 12 (OLE)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Percentage of ejected blood
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 62 | 53
Percentage of ejected blood |  |  | 3.97 (6.647) | 3.46 (5.984)

24. Secondary Outcome: Change in B-type Natriuretic Peptide (BNP) From OLE Baseline to Predefined Timepoints (OLE)
Description: BNP is small protein produced in large amounts when the heart senses it needs to work harder, such as in heart failure. Mean change from baseline (post-baseline value - OLE baseline value) in plasma BNP was calculated.
Time Frame: Baseline, Weeks 2-4, Week 8, Months 4 and 12 (OLE)
Population: FAS-Ext: The full analysis set for OLE epoch (FAS-Ext) included all subjects in the extension population who received at least one dose of the extension study drug.
  Number of participants at each post-time point (i.e., n) indicates the number of patients who have both baseline and post-time point values.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
pg/mL
  Weeks 2-4 (n = 0, 0, 78, 70): number analyzed (Participants) | 0 | 0 | 78 | 70
  Weeks 2-4 (n = 0, 0, 78, 70) |  |  | -81.78 (402.754) | 89.77 (336.742)
  Week 8 (n = 0, 0, 78, 68): number analyzed (Participants) | 0 | 0 | 78 | 68
  Week 8 (n = 0, 0, 78, 68) |  |  | -34.86 (509.893) | 170.87 (492.707)
  Month 4 (n = 0,0, 76, 69): number analyzed (Participants) | 0 | 0 | 76 | 69
  Month 4 (n = 0,0, 76, 69) |  |  | 12.86 (515.351) | 200.87 (672.071)
  Month 12 (n = 0,0, 71, 66): number analyzed (Participants) | 0 | 0 | 71 | 66
  Month 12 (n = 0,0, 71, 66) |  |  | 115.11 (600.797) | 153.06 (479.813)

25. Secondary Outcome: Change in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) From OLE Baseline to Predefined Timepoints (OLE)
Description: NT-proBNP is small protein produced in large amounts when the heart senses it needs to work harder, such as in heart failure. Mean change from baseline (post-baseline value - OLE baseline value) in plasma NT-proBNP was calculated.
Time Frame: Baseline, Weeks 2-4, Week 8, Months 4 and 12 (OLE)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
pg/mL
  Weeks 2-4 (n = 0, 0, 78, 70): number analyzed (Participants) | 0 | 0 | 78 | 70
  Weeks 2-4 (n = 0, 0, 78, 70) |  |  | -235.73 (1642.510) | -333.12 (829.689)
  Week 8 (n = 0, 0, 78, 68: number analyzed (Participants) | 0 | 0 | 78 | 68
  Week 8 (n = 0, 0, 78, 68 |  |  | -219.47 (1876.166) | -279.53 (806.447)
  Month 4 (n = 0,0, 76, 69): number analyzed (Participants) | 0 | 0 | 76 | 69
  Month 4 (n = 0,0, 76, 69) |  |  | -83.49 (798.424) | -280.35 (930.407)
  Month 12 (n = 0,0, 71, 66): number analyzed (Participants) | 0 | 0 | 71 | 66
  Month 12 (n = 0,0, 71, 66) |  |  | 266.43 (1201.239) | -358.98 (995.833)

26. Secondary Outcome: Change in Urine cGMP From OLE Baseline to Predefined Timepoints (OLE)
Description: Urinary Cyclic GMP (cGMP) is a biomarker measured in the urine that reflects the activity of biomarkers such as BNP (Brain Natriuretic Peptide). Spot urine samples were collected. Mean change from baseline (post-baseline value - OLE baseline value) in urine cGMP was calculated.
Time Frame: Weeks 2-4, Week 8, Months 4 and 12 (OLE)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
nmol/L
  Weeks 2-4 (n = 0, 0, 78, 69): number analyzed (Participants) | 0 | 0 | 78 | 69
  Weeks 2-4 (n = 0, 0, 78, 69) |  |  | 106.78 (1139.886) | 411.16 (956.355)
  Week 8 (n = 0, 0, 78, 68): number analyzed (Participants) | 0 | 0 | 78 | 68
  Week 8 (n = 0, 0, 78, 68) |  |  | 142.59 (1005.718) | 356.41 (885.854)
  Month 4 (n = 0, 0, 76, 68): number analyzed (Participants) | 0 | 0 | 76 | 68
  Month 4 (n = 0, 0, 76, 68) |  |  | 176.50 (1023.525) | 580.40 (1021.542)
  Month 12 (n = 0, 0, 71, 66): number analyzed (Participants) | 0 | 0 | 71 | 66
  Month 12 (n = 0, 0, 71, 66) |  |  | -131.86 (1284.239) | 493.21 (1024.247)

27. Secondary Outcome: Association Between Change in NT-proBNP Concentration and Change in Echocardiographic Parameters From OLE Baseline at Month 12 (OLE)
Description: Association (using the Pearson correlation coefficient) between change from OLE baseline in log-transformed NT-proBNP and echocardiographic parameters (LAVi, LVEDVi, LVESVi & LVEF)
Time Frame: Month 12
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Peason's correlation
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
Number analyzed (Participants) | 0 | 0 | 79 | 71
Peason's correlation
  NT-proBNP / LAVi( =0,0, 67, 55): number analyzed (Participants) | 0 | 0 | 67 | 55
  NT-proBNP / LAVi( =0,0, 67, 55) |  |  | 0.0178 [-0.2235 to 0.2567] | 0.0640 [-0.2054 to 0.3232]
  NT-proBNP/ LVEDVi (n = 0, 0, 62, 53): number analyzed (Participants) | 0 | 0 | 62 | 53
  NT-proBNP/ LVEDVi (n = 0, 0, 62, 53) |  |  | -0.1869 [-0.4159 to 0.0675] | -0.0059 [-0.2757 to 0.2649]
  NT-proBNP / LVESVi (n = 0, 0, 62, 53): number analyzed (Participants) | 0 | 0 | 62 | 53
  NT-proBNP / LVESVi (n = 0, 0, 62, 53) |  |  | -0.0775 [-0.3205 to 0.1762] | 0.0047 [-0.2660 to 0.2746]
  NT-proBNP / LVEF (n = 0, 0, 62, 53): number analyzed (Participants) | 0 | 0 | 62 | 53
  NT-proBNP / LVEF (n = 0, 0, 62, 53) |  |  | -0.2582 [-0.4756 to -0.0069] | 0.0233 [-0.2488 to 0.2915]

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from first dose of study treatment until end of treatment. Adverse events reported during double-blind treatment epoch (up to 41.59, 41.92 months for LCZ696 and Enalapril, respectively) were summarized. AEs during OLE epoch were summarized as well (24.80 months for LCZ696 (OLE epoch) and 24.15 months for Enalapril (OLE epoch).
Description: Adverse Event (AE): Any sign or symptom that occurs during treatment plus 30 days.
Arm/Group | LCZ696 | Enalapril | LCZ696 (Core) OLE Epoch | Enalapril (Core) OLE Epoch
All-Cause Mortality (participants affected / at risk) | 20/111 | 17/112 | 4/79 | 3/71
Serious Adverse Events (participants affected / at risk) | 64/111 | 61/112 | 38/79 | 26/71
Other Adverse Events (participants affected / at risk) | 108/111 | 108/112 | 67/79 | 64/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=111) | Enalapril (N=112) | LCZ696 (Core) OLE Epoch (N=79) | Enalapril (Core) OLE Epoch (N=71)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Acute cardiac event (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 3 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 18 | 22 | 17 | 6
Cardiac failure acute (Cardiac disorders) | 6 | 2 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 5 | 4 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 4 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 4 | 4 | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 5 | 3 | 1 | 2
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 0
Hyalosis asteroid (Eye disorders) | 1 | 0 | 0 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Large intestine polyp (Gastrointestinal disorders) | 5 | 2 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 2 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Vascular stent stenosis (General disorders) | 1 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 2 | 4 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 2
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 2 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Marasmus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 5 | 2 | 3
Embolic stroke (Nervous system disorders) | 1 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Arterial stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=111) | Enalapril (N=112) | LCZ696 (Core) OLE Epoch (N=79) | Enalapril (Core) OLE Epoch (N=71)
Anaemia (Blood and lymphatic system disorders) | 11 | 11 | 6 | 2
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 4 | 3 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 6 | 5 | 4 | 0
Atrial flutter (Cardiac disorders) | 2 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 24 | 25 | 10 | 8
Cardiac failure chronic (Cardiac disorders) | 3 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 4 | 3 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 5 | 7 | 6 | 2
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eustachian tube patulous (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 2 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 1 | 1
Thyroid disorder (Endocrine disorders) | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 0
Blepharochalasis (Eye disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 8 | 8 | 1 | 2
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 3 | 4 | 0 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 2 | 2 | 1 | 0
Dry eye (Eye disorders) | 2 | 3 | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 1 | 0
Eye discharge (Eye disorders) | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 1
Macular fibrosis (Eye disorders) | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0 | 0
Mydriasis (Eye disorders) | 1 | 0 | 0 | 0
Orbital myositis (Eye disorders) | 0 | 1 | 0 | 0
Posterior capsule opacification (Eye disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 2 | 0 | 0 | 1
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 5 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 0 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 4 | 1 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 14 | 18 | 6 | 4
Dental caries (Gastrointestinal disorders) | 2 | 5 | 2 | 3
Dental cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 17 | 4 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 6 | 3 | 2 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomach mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 3 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 2 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0
Disuse syndrome (General disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 3 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 2 | 0 | 0
Oedema peripheral (General disorders) | 5 | 3 | 3 | 1
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0
Pneumatosis (General disorders) | 1 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 7 | 8 | 3 | 1
Surgical failure (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 2 | 0 | 0 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 1 | 0 | 0
Congestive hepatopathy (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 8 | 5 | 3
Hepatic steatosis (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 8 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 4 | 0 | 2
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 2 | 1 | 0 | 2
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 2 | 0
Device related infection (Infections and infestations) | 0 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 0
Focal peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 7 | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 2 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 6 | 3 | 1 | 3
Hordeolum (Infections and infestations) | 2 | 2 | 0 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 8 | 7 | 1 | 2
Nasopharyngitis (Infections and infestations) | 53 | 53 | 19 | 18
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 2 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 4 | 5 | 1 | 2
Pharyngitis (Infections and infestations) | 4 | 2 | 0 | 4
Pneumonia (Infections and infestations) | 4 | 9 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 2 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 1 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 3 | 1 | 2
Tinea pedis (Infections and infestations) | 7 | 0 | 3 | 1
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Toxic shock syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Trichophytosis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 3 | 0 | 1
Vulval abscess (Infections and infestations) | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 10 | 3 | 4
Dental restoration failure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 1 | 3 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nasal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 5 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 2 | 0 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 3 | 1 | 0 | 0
Blood potassium increased (Investigations) | 3 | 1 | 0 | 1
Blood pressure decreased (Investigations) | 10 | 3 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure systolic decreased (Investigations) | 1 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 2 | 1 | 0 | 0
Blood uric acid decreased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 3 | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 3 | 0 | 0 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 2 | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0
Helicobacter test positive (Investigations) | 1 | 0 | 0 | 2
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1 | 1 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Lipids abnormal (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 2
Liver function test increased (Investigations) | 1 | 1 | 1 | 1
Occult blood (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Prothrombin time abnormal (Investigations) | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 1 | 0
Renal function test abnormal (Investigations) | 0 | 1 | 0 | 0
SARS-CoV-2 test negative (Investigations) | 0 | 0 | 1 | 1
Tri-iodothyronine free decreased (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 5 | 0 | 0 | 0
Weight increased (Investigations) | 4 | 4 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 2 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 17 | 8 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 10 | 5 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 4 | 3 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 17 | 5 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 6 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 5 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 9 | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 16 | 3 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 11 | 7 | 1 | 5
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 7 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 2 | 0
Monoplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0
Postresuscitation encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 2 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 3 | 2 | 3
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Eating disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Gambling disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 10 | 10 | 4 | 4
Restlessness (Psychiatric disorders) | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 2 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 2 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 18 | 23 | 11 | 6
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 2 | 0 | 3
Genital erosion (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Genital erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Combined pulmonary fibrosis and emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 7 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0 | 0
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 7 | 1 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Epidermal necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Senile pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 8 | 2 | 1
Hypotension (Vascular disorders) | 27 | 10 | 9 | 12
Internal haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 2 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the Pl to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02468232/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT02468232/SAP_001.pdf